CLINICAL TRIAL: NCT00558194
Title: Addressing Emotional and Cognitive Factors in Behavioral Weight Loss Treatment
Brief Title: Addressing Emotional and Cognitive Factors in Behavioral Weight Loss Treatment (Part 2)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funds
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23 DK73536-2; K23DK073536 (NIH)
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Overweight; Obesity
Keywords: Weight loss
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Standard behavioral weight loss treatment with cognitive and affective skills training
  Interventions: Behavioral: Standard Behavioral Weight Loss Treatment with Affective and Cognitive Skills Training
- 2 (Active Comparator): Standard behavioral weight loss treatment
  Interventions: Behavioral: Standard Behavioral Weight Loss Treatment

INTERVENTIONS:
Behavioral: Standard Behavioral Weight Loss Treatment with Affective and Cognitive Skills Training — 12-month (6-month weekly, 3-month biweekly, 3-month monthly) group treatment
  Arms: 1
Behavioral: Standard Behavioral Weight Loss Treatment — 12-month (6-month weekly, 3-month biweekly, 3-month monthly) group treatment
  Arms: 2

SUMMARY:
Behavioral weight loss, the current treatment of choice for moderate obesity, achieves impressive short term results, however, weight regain following treatment is a major problem. Over 50% of participants in behavioral weight loss programs report difficulty with internal antecedents to unhealthy weight control behaviors and this difficulty is associated with weight regain following treatment. Current treatment approaches do not adequately address these antecedents. The aim of this series of studies is to develop, implement, and evaluate a behavioral weight loss program modified to provide participants with skills to deal effectively with affective and cognitive difficulties. The study targets men and women with BMI of 27-40 who self-report difficulty with emotional and/or cognitive antecedents to unhealthy weight control behaviors. The study will randomize 120 participants to receive 12 months of standard behavioral therapy for weight loss or standard behavioral treatment plus affective and cognitive skills training. The long-term goal of this research is to improve the weight loss maintenance outcomes of behavioral weight loss programs by addressing affective and cognitive antecedents to unhealthy weight control behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 70 years
* Body mass index between 27 and 40
* Score 5 or above on the internal disinhibition scale of the Eating Inventory

Exclusion Criteria:

* Are currently participating in a weight loss program and/or are taking a weight loss medication or lost greater than or equal to 5% of body weight during the past six months
* Are pregnant, lactating, less than 6 months postpartum or plan to become pregnant during the time frame of the investigation
* Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q). Individuals endorsing joint problems, prescription medication usage, or other medical conditions that could limit exercise will be required to obtain written physician consent to participate.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Weight Loss | 12 Months

SECONDARY OUTCOMES:
Internal disinhibition as measured by the Eating Inventory | 12 Months
Physical activity as measured by the Paffenbarger | 12 months
Dietary intake as measured by the Block Food Frequency Questionnaire | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Heather M. Niemeier, Ph.D., Principal Investigator — The Miriam Hospital/The Warren Alpert Medical School of Brown U niversity
Locations (1):
- The Weight Control and Diabetes Research Center, The Miriam Hospital, Providence, Rhode Island, United States